CLINICAL TRIAL: NCT03322904
Title: Sympathetic-parasympathetic Ratio of Our Gaze
Status: Completed | Type: Observational
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Keçiören Eğitim Araştırma Hastanesi, Cardıologıst, Kecioren Education and Training Hospital
Other Study IDs: 09.03.2016/1100
Record Dates: First submitted 2017-10-10; First posted 2017-10-26 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Autonomic Nervous System Diseases
Keywords: iris collarette; autonomous nervous system
MeSH Terms: conditions — Autonomic Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: iris photography — The LF (0.04-0.15 Hz) and HF (0.16-0.4 Hz) ratings were recorded for 24 hours (day and night average) by Holter recording system
  Photographs of both irises of the healthy volunteers were taken . An image software program was used to draw circular limits over the iris exterior circle (IEC), coloretta circle (CC), and pupil circle (PC) on digital photographs. The areas between the circles were measured. The likelihood that the IRIS ratio was equal to the LF/HF ratio was calculated using the formula [IEC-PC¬] - [CC-PC] / [CC-PC].
  Other Names: holter implementation

SUMMARY:
ABSTRACT BACKGROUND The existence of the retinohypothalamic pathway suggests that light may influence autonomic outflow activity. The objective of this study was to examine the correlation between the estimated iris muscle sympathetic-parasympathetic area (IRIS) ratio and the sympathetic-parasympathetic ratio (low frequency [LF]/high frequency [HF] ratio).

METHODS The study population consisted of 200 females and 200 males (mean age, 32.4 ± 7.1 years). The IRIS ratio was determined from digital photographs of the iris in a computer setting. The LF/HF ratio was determined from records of heart rate variability obtained using a Holter implementation.

DETAILED DESCRIPTION:
INTRODUCTION The iris is the only tissue in which simultaneous interactions among smooth muscles stimulated by sympathetic and parasympathetic nerves can be observed with the naked eye. The iris contains the neural crest, which is comprised of the autonomous nervous system (ANS) and dorsal root ganglia . Fibers from the hypothalamus join the parasympathetic system through the dorsal longitudinal fasciculus and the medial forebrain bundle and unite with the Edinger-Westphal nucleus or the lateral horns of the thoracic spinal cord. A portion of these parasympathetic fibers innervate the constrictor muscle fibers of a circular structure underneath the area up to the collarette and limit the iris pupil via the oculomotor nerve. The hypothalamus is the major control and integration center of the ANS. The sympathetic nerves emerging from the hypothalamus extend along the length of the carotid artery synapse with the superior cervical ganglion and subsequently innervate the mydriasis muscle fibers beneath the iris collarette and iris root.

Heart rate variability (HRV) refers to changes in the time interval between heartbeats and is regulated by the ANS. Sympathetic and parasympathetic activities can be determined at a certain sensitivity by HRV assessment using low frequency (LF) and high frequency (HF) measurements. Previous epidemiological studies have shown that HRV is associated with both cardiac and non-cardiac all-cause mortality.

.The ANS is activated when we open our eyes, and the amount of light is adjusted by the iris . Non-visual impacts of light are mediated by melanopsin-based photoreceptors in the retinal photosensitive ganglia cells . Melanopsin is also found in the melanophores of the iris and inner brain. Phtosensitive retinal ganglion cells transmit light stimuli to the suprachiasmatic nucleus (SCN; circadian center) via the retinohypothalamic tract. In the dark, melatonin released rhythmically from the pineal gland also strongly affects SCN neuronal activity. This area receives stimulation from the visual photoreceptor system and from various areas of the brain, including the brain stem, limbic system, and cerebral cortex and contains multiple synapses with the pineal gland. The input of light into the retina, which is adjusted by the iris, is associated with the areas of the brain that regulate the ANS. Light may cause acute physiological effects such as rapid melatonin suppression, increased alertness, and increased heart rate and sympathetic nerve tonus.

The anterior cingulate cortex, amygdala, parabrachial nucleus, hypothalamus, periaqueductal grey matter, anterior insula, and some areas of the medulla play significant roles in the regulation of cardiac function. These cerebral structures are associated with cardiac activity via the sympathetic and parasympathetic nervous systems.

The objective of the study was to determine the degree of reflection of the estimated iris muscle area (IRIS) ratio of iris muscles innervated by parasympathetic and sympathetic nerves and its relationship with HRV, which is an ANS indicator of the heart.

MATERIALS AND METHODS A total of 400 healthy volunteers (200 males and 200 females) with brown eyes were included in the study. The investigators enrolled apparently healthy subjects who had no history of diabetes mellitus, hypertension, coronary artery disease, heart failure, cigarette smoking, eye disease, psychological illness, or drug therapy affecting the ANS.

A three-channel standard ambulatory Holter recording system (DMS Software Cardioscan II Holter monitoring system, ver. 11.4.0054a) was used to measure the pulse rate by HRV frequency domain analysis after removing the artefacts. The LF (0.04-0.15 Hz) and HF (0.16-0.4 Hz) ratings were recorded for 24 hours (day and night average).

Photographs of both irises of the healthy volunteers were taken using a digital camera (5-megapixel camera, 1.75 μm pixels, 0.5× digital zoom, LED flash) in the same room in daylight, at the same time of day with the same flash. Patients with non-specific and interrupted collarette (peripupillar ring) limits were not included in the study. An image software program was used to draw circular limits over the iris exterior circle (IEC), coloretta circle (CC), and pupil circle (PC) on digital photographs. The areas between the circles were measured. IEC-PC refers to the estimated total area of the dilator plus constrictor muscles stimulated sympathetically and parasympathetically; CC-PC refers to the estimated area stimulated parasympathetically; and [IEC-PC¬]-[CC-PC] refers to the estimated area stimulated sympathetically. The likelihood that the IRIS ratio was equal to the LF/HF ratio was calculated using the formula [IEC-PC¬] - [CC-PC] / [CC-PC]. The average of three measurements was calculated for each photograph.

The statistical analyses were carried out using SPSS for Windows 22 (IBM SPSS Inc., Chicago, IL, USA). The normality of the data distribution was assessed using the Kolmogorov-Smirnov test. Numerical variables with a normal distribution are presented as means ± standard deviation, while those with a nonnormal distribution are presented as medians (range). The t-test (for numerical variables displaying a normal distribution) and Mann-Whitney U-test (for numerical variables displaying an abnormal distribution) were used to determine differences between two independent groups. The association between the numerical parameters was determined by Pearson and Spearman correlation analyses. The Bland-Altman analysis was used to assess differences in compliance of the IRIS ratio and the LF/HF ratio in terms of ICC. A p-value < 0.05 was considered significant.

Studies were carried out in compliance with the Declaration of Helsinki after obtaining approval from the ethics committee. Informed consent was obtained from all subjects prior to participation.

The investigators identified a relationship between the IRIS ratio and HRV in 400 healthy subjects and demonstrated cardiac autonomic function. The IRIS ratio can also be applied to diseases accompanied by cardiac autonomic dysfunction. However, further studies are needed to demonstrate a relationship between the IRIS ratio and HRV in patients with cardiac disease.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled apparently healthy subjects

Exclusion Criteria:

* History of diabetes mellitus, hypertension, coronary artery disease, heart failure, cigarette smoking, eye disease, psychological illness, or drug therapy affecting the ANS

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 400 healthy volunteers (200 males and 200 females) with brown eyes were included in the study.
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2017-03-05 (Actual); Study Completion 2017-03-05 (Actual)

PRIMARY OUTCOMES:
Correlation between iris ratio and LF/HF ratio | 11months
  we have conducted with 400 healthly subjects iris muscle ratio associated with heart rate variability and it is demonstrated cardiac autonomic function. Iris muscle ratio can also be used in diseases accompanied by cardiac autonomic dysfunction.Correlation between pupil diameter and heart rate variability have also been investigated in some diseases where autonomic nervous system disorders are coincident. In Parkinson's disease (PD) is accompanied by autonomic nervous system dysfunction with neurodegenerative changes.. Jain et al. demonstrate simultaneous autonomic nervous system dysfunction in both pupillary diameter and in cardiac system via heart rate variability in PD Similarly, it has been shown that pupil functions in schizophrenia, which have previously been shown to be accompanied by cardiac autonomic dysfunction, may be proportional to the severity of the schizophrenia

CONTACTS AND LOCATIONS:
Overall Officials: Zuhal Koç, specialist, Study Chair — Saglik Bilimleri Universitesi
Locations (1):
- Şahbender Koç, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No